CLINICAL TRIAL: NCT01876641
Title: Phase 1/2 Study Epigenetic Modification of BRAF-mutated Metastatic Melanoma: Treatment of a Resistant Disease Using Decitabine Combined With Vemurafenib Plus Cobimetinib
Brief Title: Treatment of a Resistant Disease Using Decitabine Combined With Vemurafenib Plus Cobimetinib
Acronym: ML28604
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Mohammed M Milhem (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Mohammed M Milhem, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201304715
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Metastatic Melanoma; Melanoma; BRAF-mutated Metastatic Melanoma; V600EBRAF-mutated Metastatic Melanoma
Keywords: Metastatic melanoma; melanoma; BRAF-mutated Metastatic Melanoma; V600EBRAF-mutated metastatic melanoma; Decitabine; Vemurafenib
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; cobimetinib; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Treatment (Experimental): In Cohorts 1-4, a subcutaneous dose of decitabine will be administered three times/week over a 2 week period. Cohorts 5 and 6 will receive decitabine two times a week for 8 weeks and Cohorts 7 and 8 will receive decitabine three times a week for 8 weeks. Patients will start treatment with decitabine initially at the cohort in which they enter the study. Patients will remain in the cohort in which they were initially enrolled for the entire treatment course. Vemurafenib + Cobimetinib will be given continuously for subjects in Cohorts 5, 6, 7 and 8. Vemurafenib will be given on a 28-day cycle at the standard dose of 960 mg p.o. BID. Cobimetinib will be given on a 21-day cycle with a 7-day rest between cycles. Decitabine will be given for 2 cycles only. Each cycle will be 28 days long. Vemurafenib + Cobimetinib will be continued indefinitely until disease progression.
  Interventions: Drug: Vemurafenib + Cobimetinib, Decitabine

INTERVENTIONS:
Drug: Vemurafenib + Cobimetinib, Decitabine
  Other Names: ZELBORAF (Vemurafenib); DACOGEN (Decitabine)

SUMMARY:
The purpose of this study is to see if the combination of Vemurafenib with Decitabine plus Cobimetinib improves the low therapy response rate in subjects with malignant melanoma.

DETAILED DESCRIPTION:
The primary objective of the Phase I portion of this study is to evaluate the safety and tolerability of the proposed schedule of decitabine and Vemurafenib plus Cobimetinib in the treatment of metastatic melanoma.

ELIGIBILITY:
Inclusion criteria:

Male or female >/= 18 years old ECOG Performance Status of </= 2

Meet the following lab criteria:

Hematology Neutrophil count >1500/mm3 Platelet count >100,000/mm3 Hemoglobin >/= 9 g/dL Biochemistry AST/ALT </= 2.5 x upper limit of normal (ULN) or </= 5.0 x ULN if the transaminase elevation is due to disease involvement Serum bilirubin </= 1.5 x ULN Serum creatinine </=1.5 x ULN or estimated creatinine clearance >/= 50 ml/min by Cockcroft-Gault equation Total serum calcium (corrected for serum albumin) >/= 8.5 mg/dL or ionized calcium >/= 3.8 mg/dL Serum potassium >/= LLN Serum sodium >/= LLN Serum albumin >/= 3g/dl Baseline MUGA or ECHO must demonstrate LVEF >/= the lower limit of the institutional normal.

TSH and free T4 within normal limits, may be on thyroid hormone replacement Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first dose of study drug. Willing to use 2 methods of contraception, one being a barrier method during the study and for 3 months after last study drug dose.

Any patient with metastatic melanoma (any site) whose tumor is V600EBRAF positive, regardless of prior treatment.

Prior treatment with Vemurafenib will be allowed Must not have taken a hypomethylating agent. Must have had disease progression on or following most recent treatment regimen or on presentation for the first time with metastatic disease.

Patients with CNS disease are eligible for treatment only after their CNS disease has been directly addressed with radiation therapy.

Exclusion criteria:

Prior Decitabine for the treatment of cancer

Impaired cardiac function including any one of the following:

Screening ECG with a QTc > 460 msec confirmed by central lab prior to enrollment; congenital long QT syndrome; History of sustained ventricular tachycardia; History of ventricular fibrillation/torsades de pointes; Bradycardia defined as heart rate (hr) < 50 beats per minute; Patients with a pacemaker and hr >/= 50 beats per minute are eligible; Patients with a myocardial infarction or unstable angina within 6 mos of study entry; CHF (NYHA class III or IV); Right bundle branch block and left anterior hemiblock; Uncontrolled hypertension Concomitant use of drugs with a risk of causing torsades de pointes Concomitant use of CYP3A4, CYP1A2, or CYP2D6 substrates Unresolved diarrhea > CTCAE grade 1 Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of Vemurafenib Other concurrent severe or uncontrolled medical conditions Patients who have received prior therapies will be allowed to enroll after a wash-out period: Chemotherapy - 3 week (wk) wash-out; Oral agents - 2 wk wash-out (Except Vemurafenib, no wash-out period); Investigational agents - 3 wk wash-out; Immunotherapy - 4 wk wash-out; Palliative radiation therapy to bone/brain - 2 wk wash-out; Major radiation or surgical procedure - 3 wk wash-out Concomitant use of any anti-cancer or radiation therapy. No measurable disease Pregnant, breast-feeding women or WOCBP not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One method of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or have not been naturally postmenopausal for at least 12 consecutive months (who has had menses any time in the preceding 12 consecutive months).

Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom History of another primary malignancy within 5 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin Known positivity for HIV or hepatitis C Any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities per CTCAE 4.0 | From Day 1 - 28 of a 28 day cycle
  Toxicity will be assessed using the NIH-NCI Common Terminology Criteria for Adverse Events, version 4.0 (CTCAEv4). Toxicity will be decided after administration of one full cycle for patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milhem, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No